CLINICAL TRIAL: NCT03961074
Title: Iron Deficiency Anemia Among Chinese Pregnant Women (IRON WOMEN): a Multi-center Prospective Cohort Study
Brief Title: Iron Deficiency Anemia Among Chinese Pregnant Women: a Multi-center Prospective Cohort Study
Acronym: IRONWOMEN
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, Director, West China Hospital
Other Study IDs: IDA_2019
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Iron Deficiency Anemia of Pregnancy
Keywords: Iron Deficiency Anemia; iron supplements; Chinese pregnant women; adverse maternal outcomes; adverse neonatal outcome
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: Chinese women with iron deficiency anemia (IDA) during pregnancy.
  Interventions: Other: Iron deficiency anemia in Chinese pregnant women
- Control group: Chinese women without iron deficiency anemia (IDA) during pregnancy.

INTERVENTIONS:
Other: Iron deficiency anemia in Chinese pregnant women — Iron deficiency anemia exists in Chinese pregnant women during pregnancy
  Groups: Exposure group

SUMMARY:
Iron deficiency anemia during pregnancy, which may lead to adverse pregnancy outcomes, was a serious health problem in China. Various iron supplements used in different regions of China, however, the effects have not been well investigated. The objective of this study is to investigate the diagnosis, treatment and prognosis of iron deficiency and iron deficiency anemia in Chinese pregnant women.

DETAILED DESCRIPTION:
This is a nationwide multicenter prospective cohort study conducted in seven hospitals in China to investigate the diagnosis, treatment and prognosis of iron deficiency and iron deficiency anemia in Chinese pregnant women. This study will enroll about 6000-7000 pregnant women, who established a health record in the seven hospitals. Demographic characteristics, laboratory tests, behavior habits during pregnancy, mental status, and pregnancy outcomes will been collected. All information will collect by a pregnant women self-reported questionnaire and the electronic medical record system in hospitals at three timing points: 6-15 gestational weeks, 30-34 gestational weeks and one week after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who registered an antenatal care file at the survey hospital ;
* Signed informed consent.

Exclusion Criteria:

* Participated in any drug or nutritional clinical trial from 3 months before pregnancy to recruitment.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chinese pregnant women who established a health record at one of the survey hospital in seven cities of China.
Sampling Method: Probability Sample
Enrollment: 5551 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
adverse maternal outcomes | 40 weeks
  Including iron deficiency anemia rate, pregnancy hypertension syndrome rate, gestational diabetes mellitus rate, cesarean section rate, and other adverse maternal outcomes rate. The definition of adverse maternal outcome was according to International Glossary on Infertility and Fertility Care (2017), and the rate of adverse maternal outcome was calculated by the number of adverse maternal outcome divided by the total number of pregnant women.
adverse neonatal outcomes | 40 weeks
  Including miscarriage rate, premature birth rate, birth defect rate, low birth weight rate, and other adverse neonatal outcomes. The definitions of adverse neonatal outcomes were according to International Glossary on Infertility and Fertility Care (2017), and the rate of adverse neonatal outcomes were calculated by the number of advers neonatal outcomes divided by the total number of pregnancy or birth.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, Doctor, Study Chair — West China Hospital
Locations (7):
- China (7):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Chongqing Health center for women and Children, Chongqing, Chongqing Municipality
  - Xiamen Maternal and Child Care Hospital, Xiamen, Fujian
  - Hubei Maternal and Child Care Hospital, Wuhan, Hubei
  - Yanan University Affiliated Hospital, Yanan, Shanxi
  - The West China Second University Hospital, Chengdu, Sichuan
  - Women'S Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers with the agreement of the Coordinating Committee and the Ethics Committee.

REFERENCES:
- [Background] Haider BA, Olofin I, Wang M, Spiegelman D, Ezzati M, Fawzi WW; Nutrition Impact Model Study Group (anaemia). Anaemia, prenatal iron use, and risk of adverse pregnancy outcomes: systematic review and meta-analysis. BMJ. 2013 Jun 21;346:f3443. doi: 10.1136/bmj.f3443. PMID 23794316